CLINICAL TRIAL: NCT05709990
Title: Efficacy and Safety of High Dose Vitamin D Supplementation for Overactive Bladder Dry in Children: A Randomized Clinical Trial
Brief Title: Efficacy and Safety of High Dose Vitamin D Supplementation for Overactive Bladder Dry in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xing Liu (Other)
Responsible Party: Sponsor-Investigator, Xing Liu, Director of Urology, Children's Hospital of Chongqing Medical University, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022515
Record Dates: First submitted 2023-01-18; First posted 2023-02-02 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate; Tablets; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: The 3 groups will be treated at the same time
Who Masked: Investigator, Outcomes Assessor
Masking Description: outcome evaluators, and statisticians were blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High dose vitamin D supplementation (combined with standard urotherapy) (Experimental): These patients will receive high dose vitamin D supplementation (more than 2000IU daily) and behavioral therapy for 8 weeks
  Interventions: Drug: Vitamin D3
- Solifenacin succinate group (combined with standard urotherapy) (Active Comparator): These patients will receive solifenacin (5-10 mg daily) and behavioral therapy for 8 weeks
  Interventions: Drug: Solifenacin Succinate 5 MG Oral Tablet [Vesicare]
- standard urotherapy group (Active Comparator): These patients will receive behavioral therapy alone for 8 weeks.
  Interventions: Behavioral: Standard urotherapy

INTERVENTIONS:
Drug: Solifenacin Succinate 5 MG Oral Tablet [Vesicare] — These patients will receive solifenacin 5-10 MG daily (combined with standard urotherapy) for 8 weeks.
  Other Names: standard urotherapy
  Arms: Solifenacin succinate group (combined with standard urotherapy)
Drug: Vitamin D3 — These patients will receive high dose vitamin D supplementation (more than 2000IU daily) (combined with standard urotherapy) for 8 weeks.
  Other Names: standard urotherapy
  Arms: High dose vitamin D supplementation (combined with standard urotherapy)
Behavioral: Standard urotherapy — These patients will receive standard urotherapyfor 8 weeks.
  Arms: standard urotherapy group

SUMMARY:
This prospective, randomized, 3-arms, parallel-design, controlled clinical trial is conducted to determine whether high dose vitamin D supplementation (combined with standard urotherapy ) improves outcomes, compared with solifenacin (combined with standard urotherapy ) ,and standard urotherapy alone in children with OAB dry.

DETAILED DESCRIPTION:
Overactive bladder(OAB), characterized as urinary urgency accompanied in many instances by frequency and sometimes nocturia, with or without urinary incontinence, in the absence of urinary tract infection or other documented pathology, is a common clinical entity in pediatric urology. The majority of patients with OAB do not experience incontinence yet suffer from symptoms of urgency, frequency, and nocturia, which has been termed OAB dry. Currently, standard urotherapy is proposed as the first-line therapeutic options and adjunctive anticholinergics are usually used when urotherapy alone failed. Behavioral therapy often fail to achieve satisfied symptom control as children's poor compliance. In addition,adverse side effects such as dry mouth, constipation, gastro-oesophageal reflux result in early pharmacologic treatment discontinuation.

It was informed that patients with OAB are more likely to suffer from vitamin D deficiency. The aim of the study is to determine the effect of vitamin D supplementation as an adjunctive therapy to behavioral therapy in the treatment of OAB dry. Eligible patients aged 5-18 years with a diagnosis of OAB dry will be randomly assigned into three groups to receive high dose vitamin D supplementation (combined with standard urotherapy ) , solifenacin (combined with standard urotherapy ) or standard urotherapy alone. Serum levels of 25(OH)D will be measured at baseline. Symptoms severity will be assessed at baseline and followup. All the other sociodemographic data will be also assessed. The study will give more information on the application of vitamin D supplementation in the management of OAB dry.

ELIGIBILITY:
Inclusion Criteria:

1. Children older than 5 years of age with a diagnosis of OAB dry (do not experience incontinence yet suffer from symptoms of urgency, frequency, and nocturia) seen at the outpatient urology clinics (diagnosis follows the latest International Children's Continence Society recommendations).
2. Children with a serum vitamin D level of less than 35 ng/ml as indicated by the laboratory result.
3. Written informed consent was obtained from participants and their parents. -

Exclusion Criteria:

1. Those with a comorbidity of other urological abnormalities or serious diseases (e.g. hypospadias, cryptorchidism, posterior urethral valves, vesicoureteral reflux, neurogenic bladder, urological tumours, urinary stones, bladder and urethral injuries, etc.).
2. Those with a comorbidity of neurological disorders (e.g. epilepsy, spinal cord injury, spinal cord dysplasia, spinal cord embolism syndrome, multiple sclerosis, autism spectrum disorder, etc.) .
3. Those with acomorbidity of severe heart disease, abnormal liver or kidney function, lung disease, skeletal deformities, severe gastrointestinal disease, or inherited metabolic disorders.
4. Those with a history of gastrointestinal surgery and urinary tract surgery.
5. Those with chronic constipation.
6. Those taking anticonvulsant and antiepileptic drugs, hormones, anti-tuberculosis drugs.
7. Those have a previous history of hypercalcemia, hyperphosphatemia with renal rickets.
8. Those have a history of haematuria and urinary tract infection within the last 1 year.
9. Those have a history of allergy or allergic disease to vitamin D preparations.
10. Those Participate in other clinical studies at the time of consultation or during the follow-up of other clinical studies.
11. Any condition that could cause urinary symptoms or interfere with assessment of efficacy parameters.
12. Those unwilling to participate in this study. -

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 303 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Change in voiding frequency | 8 weeks
  Change in voiding frequency as documented in the bladder diaries (voids/d) from baseline to the followup

SECONDARY OUTCOMES:
Change in mean urgency score | 8 weeks
  Change in mean urgency score as documented from baseline to the followup，0 indicated no urgency, 1 indicated mild awareness of urgency that iseasily tolerated, 2 indicated moderate urgency discomfort that interferes with or shortens usual activity, and 3 indicated severe urgency discomfort that abruptly stops all activities or tasks
Change in max urgency score | 8 weeks
  Change in max urgency score as documented from baseline to the followup，0 indicated no urgency, 1 indicated mild awareness of urgency that iseasily tolerated, 2 indicated moderate urgency discomfort that interferes with or shortens usual activity, and 3 indicated severe urgency discomfort that abruptly stops all activities or tasks
Change in pediatric lower urinary tract symptom score | 8 weeks
  Change in pediatric lower urinary tract symptom score from baseline to the followup， score ranged from 0 to 21 and higher scores indicated a more frequent and severe occurrence of lower urinary tract symptoms.
Change in quality of life score | 8 weeks
  The quality of life was assessed using a scale ranging from 0 to 3, where a score of 0 indicated no impact on family, social, or academic life, a score of 1 indicated occasional impact, a score of 2 indicated significant impact, and a score of 3 indicated severe impact on family, social, or academic life.
Change in mean nocturia frequency, episodes/night | 8 weeks
  Change in mean nocturia frequency from baseline to the followup
Change in vitamin D level | 8 weeks
  Change in vitamin D level from baseline to the followup
Global perception of improvement | 8 weeks
  Global perception of improvement (much better; better; about the same; worse)
Wish to receive another form of treatment? | 8 weeks
  Wish to receive another form of treatment? (YES; No)

CONTACTS AND LOCATIONS:
Overall Officials: Xing Liu, Doctor, Study Director — Children's Hospital of Chongqing Medical University
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Apart from the participant's personal information.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 8 weeks
Access Criteria: Apart from the participant's personal information

REFERENCES:
- [Background] Austin PF, Bauer SB, Bower W, Chase J, Franco I, Hoebeke P, Rittig S, Vande Walle J, von Gontard A, Wright A, Yang SS, Neveus T. The standardization of terminology of lower urinary tract function in children and adolescents: update report from the Standardization Committee of the International Children's Continence Society. J Urol. 2014 Jun;191(6):1863-1865.e13. doi: 10.1016/j.juro.2014.01.110. Epub 2014 Feb 4. PMID 24508614
- [Background] Franco I. Overactive bladder in children. Nat Rev Urol. 2016 Sep;13(9):520-32. doi: 10.1038/nrurol.2016.152. Epub 2016 Aug 17. PMID 27530266
- [Background] Abrams P, Swift S. Solifenacin is effective for the treatment of OAB dry patients: a pooled analysis. Eur Urol. 2005 Sep;48(3):483-7. doi: 10.1016/j.eururo.2005.06.007. PMID 16005564
- [Background] Yuan P, Wang T, Li H, Lan R, Li M, Liu J. Systematic Review and Meta-Analysis of the Association between Vitamin D Status and Lower Urinary Tract Symptoms. J Urol. 2021 Jun;205(6):1584-1594. doi: 10.1097/JU.0000000000001441. Epub 2020 Nov 18. PMID 33207134
- [Background] Markland AD, Vaughan CP, Huang AJ, Kim E, Bubes VY, Tangpricha V, Buring JR, Lee IM, Cook NR, Manson JE, Grodstein F. Effect of Vitamin D Supplementation on Overactive Bladder and Urinary Incontinence Symptoms in Older Men: Ancillary Findings From a Randomized Trial. J Urol. 2023 Jan;209(1):243-252. doi: 10.1097/JU.0000000000002942. Epub 2022 Sep 6. PMID 36067369
- [Background] Brustad N, Yousef S, Stokholm J, Bonnelykke K, Bisgaard H, Chawes BL. Safety of High-Dose Vitamin D Supplementation Among Children Aged 0 to 6 Years: A Systematic Review and Meta-analysis. JAMA Netw Open. 2022 Apr 1;5(4):e227410. doi: 10.1001/jamanetworkopen.2022.7410. PMID 35420658

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT05709990/Prot_SAP_000.pdf